CLINICAL TRIAL: NCT01529840
Title: Norditropin Treatment in Subjects With Noonan Syndrome. Effects on Linear Growth and Final Height - Data Collection and Follow-up Visit
Brief Title: Somatropin Effect on Linear Growth and Final Height in Subjects With Noonan Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHNOO-1658; 2005-000042-37 (EudraCT Number)
Record Dates: First submitted 2012-01-02; First posted 2012-02-09 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Genetic Disorder; Noonan Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Noonan Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose 33 mcg/kg/day (Experimental)
  Interventions: Drug: somatropin
- High dose 66 mcg/kg/day (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Retrospective data collection based on data obtained from a prospective, open-label, randomised, parallel-group trial (S/GHD/004/NOO) combined with a present follow-up visit
  Arms: Low dose 33 mcg/kg/day
Drug: somatropin — Retrospective data collection based on data obtained from a prospective, open-label, randomised, parallel-group trial (S/GHD/004/NOO) combined with a present follow-up visit
  Arms: High dose 66 mcg/kg/day

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the effect of somatropin (Norditropin®) on final height in children with Noonan syndrome having being treated for up to 10 years with somatropin (Norditropin®) for the attainment of an optimal final height in the original trial S/GHD/004/NOO.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the original S/GHD/004/NOO trial or following the protocol for S/GHD/004/NOO without being randomised in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1990-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change in height SDS (Standard Deviation Score) from start of treatment to final height (referenced to normal population)

SECONDARY OUTCOMES:
Final height SDS
Change in height SDS from start of treatment to final height (referenced to Noonan population)
Height velocity
Change in height velocity
Sitting height
Number and proportion of subjects with final height SDS above -2 SDS
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Gothenburg, Sweden

REFERENCES:
- [Result] Osio D, Dahlgren J, Wikland KA, Westphal O. Improved final height with long-term growth hormone treatment in Noonan syndrome. Acta Paediatr. 2005 Sep;94(9):1232-7. doi: 10.1111/j.1651-2227.2005.tb02081.x. PMID 16203673
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com